CLINICAL TRIAL: NCT02767557
Title: A Multinational, Randomized, Phase II Study of the Combination of Nab-Paclitaxel and Gemcitabine With or Without Tocilizumab, an IL-6R Inhibitor, as First-line Treatment in Patients With Locally Advanced or Metastatic Pancreatic Cancer.
Brief Title: Study of Nab-Paclitaxel and Gemcitabine With or Without Tocilizumab in Pancreatic Cancer Patients
Acronym: PACTO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Inna Chen, MD, Staff Specialist, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GI1612
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Unresectable Pancreatic Carcinoma
MeSH Terms: interventions — tocilizumab; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab & Gemcitabine and nab-Paclitaxel (Experimental): Tocilizumab:
  8 mg/kg given I. V. on day 1 over 60 minutes every 28 day cycle.
  Gemcitabine:
  1000 mg/m² I. V. on day 1, day 8 and day 15 of every 28 day cycle.
  Nab-Paclitaxel:
  125 mg/m² I. V. on day 1, day 8 and day 15 of every 28 day cycle.
  Interventions: Drug: Tocilizumab; Drug: Gemcitabine; Drug: nab-Paclitaxel
- Gemcitabine and nab-Paclitaxel (Active Comparator): Gemcitabine:
  1000 mg/m² I. V. on day 1, day 8 and day 15 of every 28 day cycle.
  Nab-Paclitaxel:
  125 mg/m² I. V. on day 1, day 8 and day 15 of every 28 day cycle.
  Interventions: Drug: Gemcitabine; Drug: nab-Paclitaxel

INTERVENTIONS:
Drug: Tocilizumab — Intravenous infusion
  Other Names: (ACTEMRA®)
  Arms: Tocilizumab & Gemcitabine and nab-Paclitaxel
Drug: Gemcitabine — Intravenous infusion
Drug: nab-Paclitaxel — Intravenous infusion,
  Other Names: ABRAXANE®

SUMMARY:
This is a multicenter center, 2-arms prospective randomized phase II trial which evaluates whether tocilizumab with gemcitabine/nab-paclitaxel is more effective than gemcitabine/nab-paclitaxel.

DETAILED DESCRIPTION:
The development of new effective treatment strategies remains a major challenge in patients with PC. High levels of IL-6 and presence of a systemic inflammatory response in PC patients have been reported to correlate with worse survival. Preclinical PC models have clearly shown that anti-IL-6-receptor antibody tocilizumab in combination with chemotherapy reduced tumor growth, number of distant metastases and the local recurrence rate. Thus, blockade of IL-6-regulated signaling pathways represents a promising approach in combination with chemotherapy. Elevated C-reactive protein (CRP) alone or in combination with hypoalbuminaemia (Modified Glasgow Prognostic Score - mGPS) are induced by IL-6 and could feasibly represent surrogate markers for IL-6 bioactivity to stratify patients likely to gain benefit through targeting IL-6.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Histological or cytological pancreatic adenocarcinoma. Malignant unspecified tumor cells in cytological specimen are allowed after investigator assessment, mixed histology including adenosquamous carcinoma is allowed
* Male or non-pregnant, non-lactating females who are ≥18 years of age at the time of signing the informed consent form (ICF)
* Non-curable unresectable locally advanced or metastatic pancreatic carcinoma.
* A modified Glasgow Prognostic Score (mGPS) criteria of 1 or 2 assessed within 14 days of randomization as defined below:
* mGPS of 1: CRP > 10 mg/L and albumin ≥ 35 g/L
* mGPS of 2: CRP > 10 mg/L and albumin < 35 g/L
* No prior antineoplastic chemotherapy or anti-cancer drugs. Patients who have received neoadjuvant or adjuvant chemotherapy and who are diagnosed with loco regional recurrent or metastatic disease are not eligible
* ECOG/WHO Performance Status (PS) 0-1
* ≥ 4 weeks since prior major surgery, ≥ 2 weeks since prior minor surgery and ≥ 1 week since prior radiation therapy
* Measurable disease using the RECIST1.1 criteria, defined as lesions that can be measured in at least one dimension and which have not been previously irradiated. Longest diameter ≥ 20 mm with conventional techniques or ≥ 10 mm with spiral CT scan or MRI
* Fertile men and women of childbearing potential (defined as a sexually mature woman who (1) has not undergone hysterectomy [the surgical removal of the uterus] or bilateral oophorectomy [the surgical removal of both ovaries] or (2) has not been naturally postmenopausal for at least 24 consecutive months [ie, has had menses at any time during the preceding 24 consecutive months]) must use secure contraception methods as follows: intrauterine device, double-barrier contraception, as a condom and occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/cream/suppository), vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female, or complete abstinence from sexual intercourse from before 2 months entering the study until 6 months after end of chemotherapy
* Acceptable hematology parameters defined as:
* Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L
* Platelet count ≥ 100 x 10⁹/L
* Haemoglobin ≥ 5.6 mmol/L
* Acceptable liver function defined as:
* Serum bilirubin < 1.5 x upper limit of normal (ULN)
* ASAT/ALAT < 2.5 x ULN ( < 5 x ULN with known liver metastasis)
* Acceptable renal function with a creatinine clearance ≥ 50 mL/min/ (eg, using the Cockroft-Gault formula)
* Subjects must have signed and dated a BIOPAC IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care

Exclusion Criteria:

* Electrocardiogram (ECG) with significant modifications suggesting a high risk of occurrence of angina pectoris or high risk of arrhythmia.
* Other malignancies, except adequately treated basal carcinoma or squamous cell carcinoma of the skin or in-situ cervix carcinoma or incidental prostate cancer (T1a, Gleason score ≤ 6, PSA < 0.5 ng/ml), or any other tumor with a disease free survival of ≥ 5 years.
* History of serious or concurrent illness or uncontrolled medical disorder; any medical condition that might be aggravated by chemotherapy treatment or which could not be controlled; including, but not restricted to:
* Active infection requiring antibiotics within 2 weeks before the study inclusion
* Concurrent congestive heart failure NYHA ( class III - IV )
* Unstable angina pectoris, or myocardial infarction within 6 months and/or prior poorly controlled hypertension
* Inflammatory bowel disease (colitis, Crohns) or other serious gastrointestinal conditions associated with risk of perforation
* Peripheral neuropathy grade ≥ 2 according to CTCAE v 4.0
* Concomitant use of immunosuppressive or myelosuppressive medications that would in the opinion of the investigator, increase the risk of serious neutropenic complications.
* No known or suspected allergy to the investigational agents or any agents given in association with this trial.
* Pregnant or lactating women.
* Any psychological, familial, sociological, or geographical condition which does not permit protocol compliance and medical follow-up.
* Enrollment in any other clinical protocol or investigational study with an interventional agent or assessments that may interfere with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Overall survival at 6 months | Approximately up to 6 months.

SECONDARY OUTCOMES:
Performance status at 3 and 6 months assessed by investigator | Approximately up to 6 months.
Performance status at 3 and 6 months, assessed by patient | Approximately up to 6 months.
Progression free survival (PFS), defined as the time from the date of randomization until the earliest date of disease progression | Randomization to disease progression, or death due to any cause if sooner. Approximately up to 6 months.
Overall survival (OS), defined as the time from the date of randomization until death due to any cause. | Randomization until death due to any cause. Approximately up to 12 months.
Overall response rate (ORR) (ORR = CR + PR), according to RECIST 1.1.RECIST 1.1 | Approximately up to 6 months.
Disease control rate (DCR), (DCR = CR + PR + SD), according to RECIST 1.1. | Approximately up to 6 months.
Safety (Data on safety parameters) Safety and tolerability of the treatment regimens assessed by a summary of adverse events and clinical laboratory assessments. | Approximately up to 6 months.
Quality of Life (Quality of Life Questionnaire C30 (QLQ-C30) Version 3.0). | Approximately up to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Inna Chen, MD, Principal Investigator — Herlev & Gentofte Hospital; Olav Dajani, MD PhD, Principal Investigator — Oslo University Hospital
Locations (2):
- Herlev & Gentofte University Hospital, Denmark, Herlev, Denmark
- Department of Oncology, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chen IM, Johansen JS, Theile S, Silverman LM, Pelz KR, Madsen K, Dajani O, Lim KZM, Lorentzen T, Gaafer O, Koniaris LG, Ferreira AC, Neelon B, Guttridge DC, Ostrowski MC, Zimmers TA, Nielsen D. Randomized Phase II Study of Nab-Paclitaxel and Gemcitabine With or Without Tocilizumab as First-Line Treatment in Advanced Pancreatic Cancer: Survival and Cachexia. J Clin Oncol. 2025 Jun 20;43(18):2107-2118. doi: 10.1200/JCO.23.01965. Epub 2025 May 12. PMID 40354592